CLINICAL TRIAL: NCT03721159
Title: Quantification of Micro-RNA (miRNA)146-a in Subgingival Plaque Samples of Generalized Chronic Periodontitis Patients With and Without Coronary Heart Disease.
Brief Title: Quantification of Micro-RNA 146-a in Chronic Periodontitis and Coronary Heart Disease Subjects
Status: Completed | Type: Observational
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor and PhD guide, Meenakshi Ammal Dental College and Hospital
Other Study IDs: MADC/IRB-XI/2017/225
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Periodontal Diseases; Coronary Disease
Keywords: Micro-RNA; Chronic periodontitis
MeSH Terms: conditions — Periodontal Diseases; Coronary Disease; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: 30 Generalized chronic periodontitis subjects diagnosed with Coronary heart disease.
- Group II: 30 Generalized chronic periodontitis subjects without coronary heart disease.
- Group III: 30 Systemically healthy patients with no chronic periodontitis or coronary heart disease.

SUMMARY:
The expression and quantification of Micro-RNA 146-a, was analyzed in the subgingival plaque samples of generalized chronic periodontitis patients with and without coronary heart disease. The demographic variables and periodontal parameters were assessed and correlated with expression of micro-RNA 146-a. The quantification of levels of micro-RNA 146-a was done using Real time Polymerase chain reaction. ( RT-PCR)

DETAILED DESCRIPTION:
The quantification of the levels of MicroRNA 146-a was analyzed in subgingival plaque samples of generalized chronic periodontitis subjects with and without coronary heart disease and compared them with the healthy subject.A total of 90 subjects were selected for the study and assigned to 3 groups based on inclusion and exclusion criteria. Group I comprised of 30 subjects with Generalized chronic periodontitis diagnosed with coronary heart disease.Group II comprised of 30 subjects with Generalized chronic periodontitis without coronary heart disease and Group III comprised of 30 systemically healthy volunteers with no chronic periodontitis or coronary heart disease. Demographic variables such as age, weight,height,BMI and income and clinical parameters such as plaque index, bleeding on probing, probing pocket depth and clinical attachement levels were recorded. Subgingival plaque samples were collected from all the 3 groups. The collected samples were subject to further molecular analysis for micro-RNA expression and quantification using RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to participate in the study.
2. Patients within the age group of 35-65 years.
3. Should have ≥ 10 natural teeth.
4. For group I Generalized chronic periodontitis patients with coronary heart disease: Generalised chronic periodontitis is defined as those having 30% or more sites with clinical attachment loss (CAL) ≥ 3mm.
5. For group II Generalized chronic periodontitis patients without coronary heart disease.
6. Healthy controls were selected based on the following criteria: Probing pocket depth (PD) less than 4mm, bleeding on probing (BOP) at ≤15% of tooth sides, and no periodontal treatment (Scaling and root planning or periodontal surgery) within the previous six months.

Exclusion Criteria:

1. Patients with systemic conditions such as type I, type II and pre diabetes mellitus, respiratory diseases, renal disease, liver disease, collagenosis, rheumatoid arthritis, allergy, advanced malignancies and HIV infection were excluded from the present investigation.
2. Use of drugs such as corticosteroids, antibiotics within 6 month of investigation and immuno-suppressive chemotherapy.
3. Smokers and other behavioural factors which may influence the study.
4. Patients who had undergone periodontal therapy within the previous 6 months.
5. Female patients (due to hormonal changes and pregnancy which may alter the oral flora).

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients in the age group of 35-65 years were included. Females were excluded due to hormonal changes or pregnancy that may alter the oral flora
Study Population: All male patients within the age group of 35-65 years. The subjects were from South Indian population.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Micro-RNA 146-a expression in Chronic periodontitis patients with and without coronary heart disease | 9 months
  Expression of Micro-RNA 146-a using real time PCR

SECONDARY OUTCOMES:
Levels of Micro-RNA 146-a in chronic periodontitis patients with and without coronary heart disease | 9 months
  Levels of Micro-RNA 146-a using real time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Mahendra, MDS,PhD, Study Director — Meenakshi Ammal Dental College
Locations (1):
- Meenakshi Ammal Dental college, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie YF, Shu R, Jiang SY, Liu DL, Zhang XL. Comparison of microRNA profiles of human periodontal diseased and healthy gingival tissues. Int J Oral Sci. 2011 Jul;3(3):125-34. doi: 10.4248/IJOS11046. PMID 21789961